CLINICAL TRIAL: NCT01832948
Title: Study of Endostar Combined With mFOLFOX6 for First-line Treatment of Metastatic Colorectal Cancer and Efficacy Prediction
Brief Title: Endostar Combined With mFOLFOX6 for First-line Treatment of Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20121201E-mCRC
Record Dates: First submitted 2013-03-31; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — endostar protein; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Endostar d1-d7 15mg/d Oxaliplatin 85 mg/m2 d6 Folinic acid 400 mg/m2 d6 5-FU 400 mg/m2 d6, and then 5-FU 2,400 mg/m2 INTRAVENOUS over 46 h
  Interventions: Drug: Endostar; Drug: Oxaliplatin; Drug: Folinic acid; Drug: 5-FU

INTERVENTIONS:
Drug: Endostar
Drug: Oxaliplatin
Drug: Folinic acid
Drug: 5-FU

SUMMARY:
This study is to assess the efficacy and safety of Endostar combined with mFOLFOX6 in untreated metastatic colorectal cancer patients, and to find the markers that may predict the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic colorectal cancer (adenocarcinoma)
* At least one measurable lesion (RECIST criteria)
* Life expectancy ≥ 3 months
* ECOG performance status 0-2
* Adequate hematologic function: ANC ≥ 1.5×109 /L，Hb ≥ 90 g/L，PLT ≥ 100×109 /L
* Adequate renal function: Cr ≤ 1.25×ULN or Creatinine clearance ≥ 60 ml/min
* Adequate hepatic function: BIL ≤ 1.5×ULN, ALT/AST ≤ 2.5×ULN, Alkaline phosphatase ≤ 5×ULN
* Patients have not previously received palliative chemotherapy, immunological/ biological treatment
* No adjuvant chemotherapy in last six months
* Target lesion has not received local radiotherapy
* Written informed consent

Exclusion Criteria:

* Diagnosis of colorectal neuroendocrine tumor, undifferentiated carcinoma, adenosquamous carcinoma, squamous cell carcinoma
* Evidence of serious or uncontrolled infection
* Serious cardiovascular disease (congestive heart failure, uncontrollable arrhythmia, unstable angina, myocardial infarction, serious heart valve disease, resistant hypertension)
* Pregnant or lactating women
* Women of childbearing potential refused to practice acceptable methods of birth control to prevent pregnancy
* Allergic to any of the study drug
* Intestinal obstruction, intestinal perforation, or stroke within 3 months
* Participation in other clinical studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | the end of the 3rd cycle

SECONDARY OUTCOMES:
Blood perfusion in tumor tissue | baseline, the end of the 3rd cycle
Ratio of blood perfusion in tumor tissue to blood perfusion in surrounding normal tissue | baseline, the end of the 3rd cycle
Incidence of Adverse Events | up to 1 month after the last cycle

CONTACTS AND LOCATIONS:
Overall Officials: Liming Zhu, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China